CLINICAL TRIAL: NCT03981861
Title: Metabolic and Neuro-Endocrine Effect of Treating PCOS in Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16010020
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: PCOS
MeSH Terms: interventions — Metformin; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall Study (Experimental): Treatment with Metformin and Spironolactone
  Interventions: Drug: Metformin and Spironolactone

INTERVENTIONS:
Drug: Metformin and Spironolactone — Oral Metformin tablet (500 mg/tablet) twice daily for 6 months. Oral Spironolactone tablet (50 mg/tablet) once daily for 6 months.

SUMMARY:
To exam in the effect of a combination of low dose Metformin and Spironolactone on functional brain MRI, menstrual regulation and metabolism in adolescents with PCOS.

DETAILED DESCRIPTION:
Polycystic Ovarian Syndrome (PCOS) is the most common endocrinopathy in adolescent females and also one of the most complex. Patients experience an exaggerated ovarian/adrenal androgen production in response to physiologic and supra-physiologic elevations in insulin. The hormonal dysregulation is not only associated with acne, hirsutism, and menstrual irregularity, but also with perpetuated insulin resistance, central adiposity, and clinical depression.

In the proposed study, we aim to treat a hormonally and metabolically well-defined group of adolescent girls with PCOS with a combination of two pharmacological agents: metformin (insulin sensitizer) and spironolactone (anti-androgen) for 6 months. Although hyperandrogenism is a fundamental component of PCOS and responsible for the perpetuation of insulin resistance, adiposity and anovulation, there are few pediatric studies that have examined the benefits of treating both insulin resistance and hyperandrogenism simultaneously. Preliminary studies in adults, however, suggest synergistic effect of both spironolactone and metformin (spiro-met) with near normalization of the metabolic and ovulatory dysfunction. Therefore, we hypothesize that spiro-met will improve adolescent metabolism, body composition, ovarian morphology/function. We anticipate that our study will generate key pilot data for further randomized, double blind placebo controlled trials using both agents.

We also plan to examine functional brain MRI before and after the spiro-met intervention. This will allow us to inspect the effects of the hyperinsulinemic/androgenic hormonal milieu in PCOS on structural and functional brain MRI. We hypothesis, that the hormonal environment in PCOS affects centers of appetite and mood.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Meeting Androgen Excess Society (AES) diagnostic criteria of PCOS: Menstrual Dysfunction or PCO ovaries on ultrasound AND clinical or biochemical hyperandrogenism
* Normal liver and kidney function
* No chronic illnesses except for stable, treated hypothyroidism

Exclusion Criteria:

* Use of metformin and/or spironolactone within the last 6 months
* Currently on either oral hormonal contraception or other forms of hormonal contraception such as Depo-Provera, NuvaRing
* Current or past pregnancy
* Currently sexually active
* Psychiatric disorder based on self/parental report
* Type 2 diabetes (blood glucose > 200mg/dl on OGTT)
* Anemia (Hct < 35)
* Impaired kidney function (Baseline creatinine > 1.0 mg)
* Abnormal liver transaminases > 2 x the upper limit of normal range
* Potassium elevated outside the reference range (in non-hemolyzed blood sample)

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07-02 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tania Burgert, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: The pilot study was a non-controlled open label drug intervention study in a sample of adolescent girls attending a polycystic ovary syndrome (PCOS) clinic. Subjects received 6 months combination drug therapy with a combination of low dose metformin and spironolactone.
Period: Overall Study
Arm/Group | Overall Study
Started | 12
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Treatment with Metformin and Spironolactone
  Metformin and Spironolactone: Oral Metformin tablet (500 mg/tablet) twice daily for 6 months. Oral Spironolactone tablet (50 mg/tablet) once daily for 6 months.
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  North America | 12
whole body insulin sensitivity index (WBISI) [Mean (Standard Deviation); unit: μU/ml] — WBISI does not have a lot of normative data to help categorize values. However, < 4.3 is deemed insulin resistant. The lower the number the more insulin resistant.
  μU/ml | 3.67 (4.39)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 36.7 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Oral Glucose Tolerance Test
Description: Measurement of glucose and insulin at baseline and 2 hours after 75g of glucola.
Time Frame: Change Measures: Baseline & 6 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Overall Study: This was a pilot non-controlled open label drug intervention study in a sample of adolescent girls attending a polycystic ovary syndrome (PCOS) clinic. Subjects received 6 months combination drug therapy with a combination of low dose metformin and spironolactone.
Arm/Group | Overall Study
Number analyzed (Participants) | 9
mg/dL | 0.9 (2.9)

2. Primary Outcome: Total Testosterone
Description: Total Testosterone measured in ng/dL
Time Frame: Change Measures: Baseline & 6 Months
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Overall Study
Number analyzed (Participants) | 9
ng/dL | -12.57 (11.35)

3. Primary Outcome: Free Testosterone
Description: Free Testosterone measured in ng/dL
Time Frame: Change Measures: Baseline & 6 Months
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Overall Study
Number analyzed (Participants) | 9
ng/dL | -0.15 (0.24)

4. Primary Outcome: Dehydroepiandrosterone Sulfate (DHEAS)
Description: DHEAS measured in mcg/dL
Time Frame: Change Measures: Baseline & 6 Months
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Overall Study
Number analyzed (Participants) | 9
mcg/dL | -25.89 (79.07)

5. Primary Outcome: Body Mass Index (BMI)
Description: Body Mass Index measured in kg/m2
Time Frame: Change Measures: Baseline & 6 Months
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Overall Study
Number analyzed (Participants) | 9
kg/m2 | -1.3 (0.6)

ADVERSE EVENTS:
Time Frame: adverse event data was collected for the duration of the subject's intervention: 6 months
Description: Metformin is not known to cause death or hospitalization.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; Technical problems with measurement leading to unreliable or uninterpretable data. Study was not published for this reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT03981861/Prot_SAP_000.pdf